CLINICAL TRIAL: NCT03715283
Title: A Randomized Double Blind Longitudinal Study to Determine Motor Unit Number Index Variability in CMT1A Patients Undergoing a Home Ankle Strengthening Program Versus Standard of Care
Brief Title: Change in MUNIX in Patients With CMT1A Undergoing a Home Ankle Strengthening Program Versus Standard of Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Ryan Castoro, Resident Physician, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: VR52854
Record Dates: First submitted 2018-10-08; First posted 2018-10-23 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Charcot-Marie-Tooth Disease
Keywords: MUNIX
MeSH Terms: conditions — Charcot-Marie-Tooth Disease | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Lower Extremity Strengthening (Experimental): Patients in this arm will undergo a 12 week strengthening program which focuses on ankle dorsi- and plantar- flexion. Clinical visits will occur at baseline, 6 weeks and 12 weeks from the start of study. At each visit all patients will undergo a clinical exam, answer questionaires and undergo MUNIX testing.
  Interventions: Other: Home Ankle Strengthing Program
- No intervention (Experimental): In this portion of the study patients will not be given any intervention. Clinical visits will occur at baseline, 6 weeks and 12 weeks from the start of study. At each visit all patients will undergo a clinical exam, answer questionaires and undergo MUNIX testing of both legs.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Home Ankle Strengthing Program — Patients in this arm will be given a USB or DVD video with description of ankle dorsi- and plantar- flexion resistance band exercise. They will also be given an outlined plan for there exercises, progression and an exercise diary. In general patients will start with a low resistance and low reps, over the 4 weeks they will increase the repetitions at the same resistance band. After the 4 weeks they will have the option to escalate the band resistance or continue at the same resistance and repetitions until comfortable progressing. The same 4 week progression will be used for each resistance band over the 12 weeks.
  Arms: Home Lower Extremity Strengthening
Other: Standard of Care — Patients in this arm will be directed to continue there standard care program. They will be asked to refrain from resistance exercise for 12 weeks.
  Arms: No intervention

SUMMARY:
Here the investigators aim to show that a focused lower extremity resistance strength training program in patients with Charcot-Marie-Tooth disease (CMT) results in increased motor strength of ankle plantar- and dorsi-flexion. The investigators will use motor unit index MUNIX and hand held dynamometry to correlate strength changes. The investigators believe that increased strength will correlate with an increased motor unit number and as such will prove that axonal renervation or improved recruitment is possible with a focused exercises in patients with CMT. Additionally, the investigators will show that that MUNIX declines over a 12-week period in patients with CMT whom continue standard of care. This will identify MUNIX as a responsive marker for disease progression in addition to detecting functional improvement, which will be valuable for future clinical trials.

DETAILED DESCRIPTION:
1. Overview Previous data in CMT patients on strengthening programs have had mixed results. No studies have demonstrated the effectiveness of a home exercise resistance band training program on ankle dorsiflexion strength in CMT patients. Additionally, it has been shown that that MUNIX is associated with disability scores and could be used as an outcome measure in CMT. Here the investigators will perform a randomized clinical trial to assess the ability of MUNIX to detect longitudinal changes in patients with CMT undergoing an ankle strengthening program.
2. AIM 1: To determine if adult patients with CMT1A whom undergo a twelve-week ankle strengthening program will have a significant increase in ankle dorsi- and plantar- flexion, as measured by muscle strength dynamometry compared to patients whom do not undergo the program. Patients enrolled in this study will be randomized to receive either a 12-week home resistance band ankle strengthening program or to continue their current treatment plan. Clinical evaluations and 6-minute walk test will be performed in all enrolled patients, regardless of their arm, at the time of enrollment, 6 and 12 weeks after enrollment. A parallel study of healthy unaffected family members will also be performed in this basis.
3. Resistance Band Strengthening Exercises Patients assigned to the strength training group will be a given a twelve-week progressive resistance band program. Study materials in the treatment arm will include a written exercise plan accompanied by a USB and DVD containing demonstration of safe execution of each exercise. Patients in the treatment arm will perform each exercise three times per week. A All exercises are meant to be performed in a seated or lying position for safety.
4. Clinical evaluations The investigators will perform all clinical assessments at the Vanderbilt Physical Medicine and Rehabilitation clinic and will be performed by the PI. To maintain blinding by the PI, a pre-determined set of questions will be asked of each patient in order to prevent inadvertent unblinding. Examples of the questionnaires for the 6 and 12 weeks follow up visits are found in the study materials section.

   . History taking and Neurological examination
   * Medical history: The patient will be interviewed by the PI to collect medical history, particularly for symptoms relating the peripheral nerves and family history.
   * Neurological examination: Each patient will be examined by the PI. Findings on neurological examination will be recorded, particularly for the sensory and motor functions.

     * The Motor portion of the exam will be performed by hand held digital dynamometry as has been previously described
     * For the Sensory portion of the exam the investigators will test pinprick, vibratory and light sensations bilaterally
   * CMT neuropathy score (CMTNS): This is a simple, extensively validated(16), score system that assesses the disabilities in a patient with CMT. It consists of a brief questionnaire, physical findings and several parameters from nerve conduction studies. For the purposes of this study only the symptom score and examination score. An example of the modified CMTNS is provided in the study materials section.
5. 6-minute walk test The six-minute walk test (6MWT) will be performed at the enrollment visit, 6 and 12 weeks after enrollment. This will be performed in the Physical Medicine and Rehabilitation clinic at Vanderbilt University Medical Center. Testing will be conducted as outlined by the American Thoracic Society with some modifications.

   For the purposes of this study a 10m hallway will be marked with cones. The patient will walk for 6 minutes and forth along the marked hallway. The patient may rest during the 6 minutes. The total distance walked, and number of rest breaks will be recorded. Patients whom use assistive devices such as walkers, canes or ankle braces may will not be asked to undergo the walk if a participant does not feel comfortable ambulating without a device. The PI will accompany each patient with a wheelchair during the entire 6 minutes in case an immediate break is needed. If participants are unable to participate in the 6MWT at the initial visit, participants will be excluded from this portion of the study due to risk of unblinding, but will continue in the study.

   The 6MWT is contraindicated in patients with unstable angina and those whom have had a myocardial infarction within the last month. Any patient with a positive history will not undergo testing. Each patient will have their seated pulse and blood pressure checked prior to the test. Patients with a pulse rate of 120 beats per minute or greater or a systolic blood pressure greater than 180mmHg (mmHg = millimeter of Mercury) or diastolic blood pressure of 100mmHg or greater will not undergo testing. If elevated blood pressure or pulse is found at the initial clinical encounter, the patient's primary physician will be contacted, and the patient will be brought back at least 2 weeks but no more than 3 weeks later for a blood pressure and pulse check. If the blood pressure or pulse is within the limits defined above, participants will be allowed to undergo testing at this later date. If participants continue to have elevated blood pressure or pulse, participants will not undergo this portion of the study.
6. AIM2: MUNIX Studies Procedural and interpretative guidelines for MUNIX have recently been published and will followed in this study. Here the investigators will study the tibialis anterior and abductor hallucis. The tibialis anterior is innervated by deep peroneal branch of the peroneal nerve. Whereas the abductor hallucis is innervated by the tibial nerve. Each muscle will be studied in the extremity with best strength in both ankle dorsiflexion and plantar flexion. If there is a difference between the two muscles the limb with best ankle dorsiflexion strength will be used. All studies will be performed in the VUMC Electrodiagnostic laboratory by the PI.

Prior to the start of the study, lower extremity surface temperature will be measured in the on the lateral aspect of the lower leg that is being tested. If patients surface temperature is below 32oC (or if temperature falls below during the study), a warming pad or heating lamp will be applied. Then at each recording site a supramaximal compound motor unit action potential (CMAP) will be recorded by providing an electrical stimulus over the nerve proximal to the recording sites. There will be at least 3 small adjustments of the recording electrodes to achieve maximal recording of the CMAP. Patients with no response in the CMAP will continue in the study but will be censored from initial analysis such to not askew the data.

Next surface electromyography will be performed by recording the surface interference pattern from the recording site of maximal CMAP. Patients will then perform isometric muscle contractions at 20, 40, 60, 80 and 100% of maximal effort. Following maximal effort patients will be given a 10 second rest period. This will be repeated a total of three times for each nerve tested. The MUNIX will be calculated by a propriety software from Natus (Middleton, WI). As part of the MUNIX output the motor unit size index (MUSIX) will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients 18 years or older with genetically confirmed CMT1A
* Adult Patients 18 years or older with a CMT1A genetically confirmed relative and a positive clinical exam or nerve conduction study consistent with CMT1A.
* Unaffected persons 18 years or older with no past medical history of peripheral neuropathy

Exclusion Criteria:

* Patients with a history of medical diseases that affect peripheral nerve function including diabetic neuropathy, uncontrolled thyroid dysfunction, amyloidosis, monoclonal gammopathy of uncertain significance or untreated vitamin deficiencies.
* Patients with a history of other neurologic disease which may affect peripheral nerve function or extremity strength or function including stroke, seizures with a history of Todd's paralysis, Parkinson's Disease, Dementia, Guillen-Barre Syndrome, Myasthenia Gravis, Lambert Eaton Myasthenia Gravis or hypothyroidism.
* Patients with ankle dorsiflexion strength of less than 3/5 in either limb on Medical Research Council scale.
* Patients enrolled in a clinical trial (excluding natural history studies) in the past 12 months.
* Patients who have undergone intense physical therapy, meaning more than 1 time per week for 6 or more weeks within the last 12 months.
* Patient who do resistance training of the lower extremity more than 2 times per week for more than 3 months.
* Patient in whom exercise would be consider dangerous including autonomic failure, postural orthostatic tachycardic syndrome (POTS), lower extremity deep vein thrombosis or pulmonary embolism, arterial insufficiency, uncontrolled pulmonary hypertension, uncontrolled hypertension or uncontrolled heart failure with reduced ejection fraction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Change in motor unit number index (MUNIX) of the peroneal nerve in the treatment arm versus the untreated arm from baseline to 12 weeks (Peroneal Munix at 12 weeks - Peroneal Munix at baseline,0-1,000a.u., higher numbers represent more motor units) | 12 weeks
Change in motor unit number index (MUNIX) of the tibial nerve in the treatment arm versus the untreated arm from baseline to 12 weeks (Tibial MUNIX.at 12 weeks - Tibial MUNIX at baseline, 0-1000 arbitrary units, higher numbers represent more motor units) | 12 weeks

SECONDARY OUTCOMES:
Change in peroneal nerve motor unit number index (MUNIX) at 6 weeks between treatment arms (MUNIX at 6 weeks - MUNIX at Baseline; 0-1000 arbitrary units, higher numbers represent more motor units). | 6 weeks
Change in tibial nerve compound muscle action potential (CMAP) at 6 weeks between treatment arms ((Tibial CMAP at 6 weeks - Tibial CMAP at baseline (mV) 0-300mV, mV= milliVolts, higher numbers represent more motor units). | 6 weeks
Change in tibial nerve compound muscle action potential (CMAP) at 12 weeks between treatment arms (Tibial CMAP at 12 weeks - Tibial CMAP at baseline (mV) 0-300mV, mV= milliVolts, higher numbers represent more motor units). | 12 weeks
Change in peroneal nerve compound muscle action potential (CMAP) at 6 weeks between treatment arms (Peroneal CMAP at 6 weeks - Peroneal CMAP at baseline 0-300mV, mV = milliVolts, higher numbers represent more motor units). | 6 weeks
Change in peroneal nerve compound muscle action potential (CMAP) at 12 weeks between treatment arms (Peroneal CMAP at 12 weeks - Peroneal CMAP at baseline 0-300mV, mV= milliVolts, higher numbers represent more motor units). | 12 weeks
Change in muscle strength as measured by dynamometry of ankle dorsiflexion at 6 weeks between treatment arms (dorsiflexion strength at 6 weeks - dorsiflexion strength at baseline 0- 500 N, N=Newton, higher numbers represent means greater strength). | 6 weeks
Change in muscle strength as measured by dynamometry of ankle dorsiflexion at 12 weeks between treatment arms (dorsiflexion strength at 12 weeks - dorsiflexion strength at baseline 0-500 N, N=Newton, higher numbers represent means greater strength). | 12weeks
Change in muscle strength as measured by dynamometry of ankle plantarflexion at 6 weeks between treatment arms (plantarflexion strength at 6 weeks - plantarflexion strength at baseline 0-500N, N= Newton, higher numbers represent means greater strength). | 6 weeks
Change in muscle strength as measured by dynamometry of ankle plantarflexion at 12 weeks between treatment arms (plantarflexion strength at 12 weeks - plantarflexion strength at baseline 0-500N, N= newton higher numbers represent means greater strength). | 12 weeks
Change in the 6 minute walk test (6MWT) at 6 weeks between treatment arms (6MWT at 6 weeks - 6MWT at baseline 0-5,000m; m = meter, longer distances represent improved functional mobility). | 6 weeks
Change in the 6 minute walk test (6MWT) at 12 weeks between treatment arms (6MWT at 12 weeks - 6MWT at baseline 0-5,000m; m = meter, longer distances represent improved functional mobility). | 12 weeks
Change in Charcot Marie Tooth Disease neuropathy score (CMTNS) at 12 weeks between treatment arms (CMTNS at 12 weeks - CMTNS at baseline 0-36 arbitrary units, higher numbers represent more severe disease). | 12 weeks
Change in Charcot Marie Tooth Disease neuropathy score (CMTNS) at 6 weeks between treatment arms (CMTNS at 6 weeks - CMTNS at baseline 0-36 arbitrary units, higher numbers represent more severe disease). | 6 weeks
Change in peroneal nerve motor unit size index (MUSIX) at 6 weeks between treatment arms (Peroneal MUSIX at 6 weeks - Peroneal MUSIX at Baseline 0-1,000 arbitrary units, higher number represents more motor units). | 6 weeks
Change in peroneal nerve motor unit size index (MUSIX) at 12 weeks between treatment arms (Peroneal MUSIX at 12 weeks - Peroneal MUSIX at Baseline 0-1,000 arbitrary units, higher number represents more motor units). | 12 weeks
Change in tibial nerve motor unit size index (MUSIX) at 6 weeks between treatment arms (Tibial MUSIX at 6 weeks - Tibial MUSIX at Baseline 0-1,000 arbitrary units, higher number represents more motor units). | 6 weeks
Change in tibial nerve motor unit size index (MUSIX) at 12 weeks between treatment arms (Tibial MUSIX at 12 weeks - Tibial MUSIX at Baseline 0-1,000 arbitrary units, higher number represents more motor units). | 12 weeks
Change in tibial nerve motor unit number index (MUNIX) at 6 weeks between treatment arms (MUNIX at 6 weeks - MUNIX at Baseline; 0-1000 arbitrary units, higher number represents more motor units). | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Castoro, D.O., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li J. Inherited neuropathies. Semin Neurol. 2012 Jul;32(3):204-14. doi: 10.1055/s-0032-1329198. Epub 2012 Nov 1. PMID 23117945
- [Background] Nandedkar SD, Barkhaus PE, Stalberg EV. Motor unit number index (MUNIX): principle, method, and findings in healthy subjects and in patients with motor neuron disease. Muscle Nerve. 2010 Nov;42(5):798-807. doi: 10.1002/mus.21824. PMID 20976783
- [Background] Bas J, Delmont E, Fatehi F, Salort-Campana E, Verschueren A, Pouget J, Lefebvre MN, Grapperon AM, Attarian S. Motor unit number index correlates with disability in Charcot-Marie-Tooth disease. Clin Neurophysiol. 2018 Jul;129(7):1390-1396. doi: 10.1016/j.clinph.2018.04.359. Epub 2018 Apr 16. PMID 29729594